CLINICAL TRIAL: NCT01626456
Title: A Phase 3, Multicenter, Extension of Study ALK9072-003 to Assess the Long-term Safety and Durability of Effect of ALKS 9072 in Subjects With Stable Schizophrenia
Brief Title: A Long-term Safety Study of ALKS 9072 (Also Known as ALKS 9070)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK9072-003EXT
Record Dates: First submitted 2012-06-15; First posted 2012-06-22 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 9072, Low (Experimental)
  Interventions: Drug: ALKS 9072, Low
- ALKS 9072, High (Experimental)
  Interventions: Drug: ALKS 9072, High

INTERVENTIONS:
Drug: ALKS 9072, Low — IM injection, given monthly
  Arms: ALKS 9072, Low
Drug: ALKS 9072, High — IM injection, given monthly
  Arms: ALKS 9072, High

SUMMARY:
This study will evaluate the safety and durability of effect of ALKS 9072 (also known as ALKS 9070) during long-term treatment of subjects with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

(Subjects who participated in ALK9072-003)

* Completed the ALK9072-003 Day 85 visit
* Continues to require treatment with an antipsychotic medication

(New Subjects)

* On a stable dose of oral antipsychotic medication
* Diagnosis of chronic schizophrenia based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria that is clinically stable
* Has been able to achieve outpatient status for more than 3 months prior to screening
* Body Mass Index (BMI) of 18.5 to 40.0 kg/m2 (inclusive)
* Resides in a stable living situation

Exclusion Criteria:

(Subjects who participated in ALK9072-003)

* Abnormal clinical laboratory, vital sign, or electrocardiogram (ECG) finding during participation in study ALK9072-003 that was clinically relevant and related to study drug
* Missed more than 1 scheduled study visit during participation in study ALK9072-003
* Has a significant or unstable medical condition that would preclude safe completion of the current study
* Subject is pregnant or breastfeeding
* Subject expects to be incarcerated in the next 12 months, or has pending legal action which may impact compliance with study participation or procedures

(New Subjects)

* History of poor or inadequate clinical response to treatment with aripiprazole
* History of treatment resistance
* Diagnosis of current substance dependence (including alcohol)
* Pregnant, lactating, or breastfeeding
* Has received any long-acting intramuscular antipsychotic medication within 60 days prior to screening
* Currently under involuntary hospitalization
* Current or expected incarceration

Additional inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (78):
- United States (21):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, La Habra, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Fort Lauderdale, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Overland Park, Kansas
  - Alkermes Investigational Site, Rockville, Maryland
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
- Bulgaria (13):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Pazardzhik
  - Alkermes Investigational Site, Pleven
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Radnevo
  - Alkermes Investigational Site, Rousse
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Stara Zagora
  - Alkermes Investigational Site, Targovishte
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Malaysia (4):
  - Alkermes Investigational Site, Cheras
  - Alkermes Investigational Site, Johor Bahru
  - Alkermes Investigational Site, Kuala Lumpur
  - Alkermes Investigational Site, Kuching
- Philippines (6):
  - Alkermes Investigational Site, Mariveles, Bataan
  - Alkermes Investigational Site, Cebu City
  - Alkermes Investigational Site, Iloilo City
  - Alkermes Investigational Site, Mandaluyong
  - Alkermes Investigational Site, Manila
  - Alkermes Investigational Site, Pasig
- Romania (5):
  - Alkermes Investigational Site, Târgu Mureş, Mureș County
  - Alkermes Investigational Site, Bucharest
  - Alkermes Investigational Site, Craiova
  - Alkermes Investigational Site, Iași
  - Alkermes Investigational Site, Oradea
- Russia (14):
  - Alkermes Investigational Site, Nikol’skoye, Gatchinckiy
  - Alkermes Investigational Site, Staritsa, Orenburg Oblast
  - Alkermes Investigational Site, Khot'kovo
  - Alkermes Investigational Site, Lipetsk
  - Alkermes Investigational Site, Moscow
  - Alkermes Investigational Site, Nizhny Novgorod
  - Alkermes Investigational Site, Rostov-on-Don
  - Alkermes Investigational Site, Saint Petersburg
  - Alkermes Investigational Site, Samara
  - Alkermes Investigational Site, Saratov
  - Alkermes Investigational Site, Stavropol
  - Alkermes Investigational Site, Talagi
  - Alkermes Investigational Site, Voronezh
  - Alkermes Investigational Site, Yaroslavl
- South Korea (3):
  - Alkermes Investigational Site, Jeju City
  - Alkermes Investigational Site, Jeollanam-do
  - Alkermes Investigational Site, Seoul
- Ukraine (12):
  - Alkermes Investigational Site, Stepanivka, Kherson Oblast
  - Alkermes Investigational Site, Chernihiv
  - Alkermes Investigational Site, Donetsk
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kyiv
  - Alkermes Investigational Site, Luhansk
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Poltava
  - Alkermes Investigational Site, Simferopol
  - Alkermes Investigational Site, Ternopil
  - Alkermes Investigational Site, Uzhhorod
  - Alkermes Investigational Site, Vinnytsia

REFERENCES:
- [Result] Hard ML, Mills RJ, Sadler BM, Turncliff RZ, Citrome L. Aripiprazole Lauroxil: Pharmacokinetic Profile of This Long-Acting Injectable Antipsychotic in Persons With Schizophrenia. J Clin Psychopharmacol. 2017 Jun;37(3):289-295. doi: 10.1097/JCP.0000000000000691. PMID 28350572
- [Derived] McEvoy JP, Weiden PJ, Lysaker PH, Sun X, O'Sullivan AK. Long-term effect of aripiprazole lauroxil on health-related quality of life in patients with schizophrenia. BMC Psychiatry. 2021 Mar 24;21(1):164. doi: 10.1186/s12888-021-03124-2. PMID 33761928
- [Derived] Lauriello J, Claxton A, Du Y, Weiden PJ. Beyond 52-Week Long-Term Safety: Long-Term Outcomes of Aripiprazole Lauroxil for Patients With Schizophrenia Continuing in an Extension Study. J Clin Psychiatry. 2020 Aug 18;81(5):19m12835. doi: 10.4088/JCP.19m12835. PMID 32841554
- [Derived] Nasrallah HA, Aquila R, Du Y, Stanford AD, Claxton A, Weiden PJ. Long-term safety and tolerability of aripiprazole lauroxil in patients with schizophrenia. CNS Spectr. 2019 Aug;24(4):395-403. doi: 10.1017/S1092852918001104. Epub 2018 Aug 15. PMID 30109845
- [Derived] Weiden PJ, Du Y, Liu CC, Stanford AD. Switching stable patients with schizophrenia from their oral antipsychotics to aripiprazole lauroxil: a post hoc safety analysis of the initial 12-week crossover period. CNS Spectr. 2019 Aug;24(4):419-425. doi: 10.1017/S1092852918000986. Epub 2018 Jun 26. PMID 29941057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who successfully completed the Day 85 visit in Study ALK9072-003 and continued to meet eligibility criteria were eligible to enroll in this extension study. In addition, adults with chronic stable schizophrenia on a stable oral antipsychotic medication not previously enrolled in Study ALK9072-003 were also eligible to enroll.
Pre-assignment Details: While there were only 2 treatment groups in this extension study (low dose and high dose), data for several outcome measures is presented by lead-in study groups, and separated into 5 categories: PBO-441 mg, 441-441 mg, PBO-882 mg, 882-882 mg, and de novo.
Period: Overall Study
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Started | 110 | 368
Completed | 75 | 251
Not Completed | 35 | 117
Not completed — Withdrawal by Subject | 21 | 46
Not completed — Adverse Event | 2 | 27
Not completed — Lost to Follow-up | 2 | 27
Not completed — Lack of Efficacy | 6 | 7
Not completed — Physician Decision | 1 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Site Closure | 2 | 3
Not completed — Incarceration | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population includes all subjects who receive at least 1 dose of ALKS 9072 in the current study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 9072, Low | ALKS 9072, High | Total
Number analyzed (Participants) | 110 | 368 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.88) | 39.8 (11.76) | 39.4 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 158 | 203
  Male | 65 | 210 | 275
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 59 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 13 | 79 | 92
  White | 77 | 228 | 305
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 20 | 60 | 80
  Romania | 3 | 2 | 5
  United States | 19 | 111 | 130
  Philippines | 17 | 32 | 49
  Ukraine | 29 | 93 | 122
  Korea, Republic of | 0 | 6 | 6
  Malaysia | 3 | 21 | 24
  Bulgaria | 19 | 43 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: This measure includes incidences >5%.
Time Frame: 52 weeks
Population: Safety population includes all subjects who receive at least 1 dose of ALKS 9072 in the current study.
Measure: Number; unit: participants
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Number analyzed (Participants) | 110 | 368
participants | 51 | 190

2. Secondary Outcome: Mean Change From Baseline to Endpoint in Clinical Global Impression Scale for Severity (CGI-S)
Description: The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is in a specific point in time. Results indicate participants evaluated at one of the following categories: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients". Results indicate a change in CGI-S score from baseline to Day 365 based on the observed data.
Time Frame: 52 weeks
Population: The full analysis set consists of all subjects who received at least 1 dose of ALKS 9072 and had at least 1 postbaseline assessment of PANSS score after administration of ALKS 9072.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PBO-441 mg: Subjects who received placebo in the base study and low dose in the current study.
- 441-441 mg: Subjects who received low dose in both the base study and the current study.
- PBO-882 mg: Subjects who received placebo in the base study and high dose in the current study.
- 882-882 mg: Subjects who received high dose in both the base study and the current study.
- De Novo: Subjects who did not participate in the base study. These subjects received high dose.
Arm/Group | PBO-441 mg | 441-441 mg | PBO-882 mg | 882-882 mg | De Novo
Number analyzed (Participants) | 29 | 80 | 26 | 94 | 233
units on a scale | -0.9 (0.68) | -0.5 (0.71) | -0.8 (0.85) | -0.3 (0.61) | -0.2 (0.61)

3. Secondary Outcome: Discontinuation From Study Due to Adverse Events (AEs)
Description: Number of subjects who discontinued the study due to AE.
Time Frame: 52 weeks
Population: Safety population includes all subjects who received at least 1 dose of ALKS 9072 in the current study.
Measure: Number; unit: participants
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Number analyzed (Participants) | 110 | 368
participants | 2 | 27

4. Secondary Outcome: Suicidal Ideation and Behavior Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a questionnaire used for suicide assessment. Subjects are asked a series of questions that determine whether or not the patient demonstrates any suicidal ideation or behavior. The C-SSRS was administered to subjects at each study visit.
Time Frame: 52 weeks
Population: Safety population includes all subjects who received at least 1 dose of ALKS 9072 in the current study.
Measure: Number; unit: participants
Groups:
- PBO-440 mg: Subjects who received placebo in the base study and low dose in the current study
- 441-441 mg: Subjects who received low dose in the base study and in the current study.
- 882-882 mg: Subjects who received high dose in the base study and the current study.
- De Novo: Subjects who did not participate in the base study.
Arm/Group | PBO-440 mg | 441-441 mg | PBO-882 mg | 882-882 mg | De Novo
Number analyzed (Participants) | 29 | 81 | 26 | 100 | 242
participants
  Any suicidal ideation | 0 | 1 | 1 | 1 | 4
  Any suicidal behavior | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Incidence of Clinically Significant Changes Will be Calculated for Movement Disorders, Vital Signs and Routine Laboratory Tests
Description: Includes incidence >2% but <5%.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | PBO-441 mg | 441-441 mg | PBO-882 mg | 882-882 mg | De Novo
Number analyzed (Participants) | 29 | 81 | 26 | 100 | 242
participants
  Akathisia | 1 | 0 | 2 | 3 | 12
  Tremor | 1 | 0 | 0 | 4 | 7
  Glycosylated haemoglobin increased | 0 | 3 | 0 | 0 | 3
  Hypertension | 1 | 0 | 1 | 3 | 4

6. Secondary Outcome: Mean Change From Baseline to Endpoint Using the Positive and Negative Symptom Scale (PANSS) Total Score and Subscale Scores
Description: This scale consists of symptom constructs (7 positive, 7 negative, 16 general psychopathology), each to be rated on a 7-point Likert-type scale of severity with 1 being absent to 7 being extreme. Minimum scores (best outcome) equals 30 (total scale), 7 (positive/negative subscales), and 16 (general subscale); maximum scores (worst outcome) equals 210 (total scale), 49 (positive/negative subscales), and 112 (general subscale).
Time Frame: 52 weeks
Population: The full analysis set consisted of all subjects who received at least 1 dose of ALKS 9072 and had at least 1 postbaseline assessment of PANSS total score after administration of ALKS 9072.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBO-441 mg | 441-441 mg | PBO-882 mg | 882-882 mg | De Novo
Number analyzed (Participants) | 29 | 80 | 26 | 94 | 233
units on a scale
  Total Score | -19.1 (15.5) | -10.0 (10.2) | -11.6 (11.7) | -8.3 (8.2) | -5.9 (8.3)
  Positive Subscale Score | -5.8 (6.0) | -3.4 (3.4) | -4.1 (4.1) | -2.3 (3.1) | -1.8 (2.8)
  Negative Subscale Score | -4.1 (4.2) | -1.5 (3.5) | -1.6 (3.8) | -2.1 (3.0) | -1.2 (3.3)
  General Psychopathology Subscale Score | -9.2 (7.6) | -5.1 (5.6) | -5.9 (6.1) | -4.0 (4.7) | -2.9 (4.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every study visit for 1 year (365 days).
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Serious Adverse Events (participants affected / at risk) | 0/110 | 15/368
Other Adverse Events (participants affected / at risk) | 16/110 | 59/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 9072, Low (N=110) | ALKS 9072, High (N=368)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 2 (2)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 9072, Low (N=110) | ALKS 9072, High (N=368)
Weight increased (Investigations) | 7 (8) | 17 (17)
Headache (Nervous system disorders) | 7 (10) | 11 (15)
Insomnia (Psychiatric disorders) | 3 (4) | 37 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/ publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.